CLINICAL TRIAL: NCT06510504
Title: A Phase 3, Randomized, Double-blind, 2-arm, Parallel-group, Placebo-controlled Study to Evaluate the Efficacy and Safety of BNC210 for the Acute, As-needed Treatment of Anxiety in Adults With Social Anxiety Disorder
Brief Title: Efficacy of BNC210 in Acute, As-needed Treatment of Anxiety in Social Anxiety Disorder - 1
Acronym: AFFIRM-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bionomics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNC210.014
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-09

CONDITIONS: Social Anxiety Disorder
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 225 mg BNC210 (Experimental)
  Interventions: Drug: 225 mg BNC210
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 225 mg BNC210 — 225 mg BNC210
  Arms: 225 mg BNC210
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effect of a single, acute dose of BNC210 compared to placebo on reducing the severity of anxiety provoked by a behavioral assessment task and measured using the Subjective Units of Distress Scale (SUDS) in adult patients with social anxiety disorder.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, 2-arm, parallel-group, multi-center study. Participants will attend a Screening Visit to confirm eligibility and then return to the clinic within 21 days to be randomized into the study. Randomized participants will receive a single dose of their allocated study medication (225 mg BNC210 or placebo) and approximately 1 hour later participate in a behavioral assessment task. After 1 week, a safety follow-up assessment will be conducted by phone/video conference.

ELIGIBILITY:
Inclusion Criteria:

* A current diagnosis of social anxiety disorder as defined in the DSM-5.
* A Liebowitz Social Anxiety Scale total score of ≥60.
* Suitable contraception use in line with protocol requirements.
* Ability to swallow tablets.

Exclusion Criteria:

* History of bipolar disorder, schizophrenia, schizoaffective disorder, psychotic disorders, anorexia or bulimia, body dysmorphic disorder, PTSD, autism-spectrum disorder or obsessive-compulsive disorder, or any other Axis I or II disorder which is currently the primary focus of treatment over social anxiety disorder.
* Hamilton Rating Scale for Depression score of ≥18.
* Moderate or severe alcohol-use disorder, or any other substance-use disorder (any severity) in the past 12 months.
* Use of psychotropic medications within 30 days of screening. Daily use of benzodiazepines within 90 days of screening.
* Any clinically significant medical history or findings as determined by the Investigator that could interfere with the objectives of the study or put the participant at risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-09-11 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Subjective Units of Distress Scale (SUDS) | 1 day
  The Subjective Units of Distress Scale (SUDS) is a self reported measure of the intensity of distress currently experienced by an individual. The range is 0-100, with a higher score indicating a higher level of anxiety/greater distress.

SECONDARY OUTCOMES:
Clinical Global Impressions-Severity (CGI-S) | 1 day
  The CGI-S measures overall disease severity of the participant's symptoms as scored by a clinician. Severity is rated from 1 (normal, not at all ill) to 7 (among the most extremely ill of patients) with a higher score indicating a higher level of disease severity.
Patient Global Impressions-Improvement (PGI-I) | 1 day
  The PGI-I is a patient self-reported counterpart of the CGI designed to assess the patient's impression of their perceived change in overall symptoms. Improvement is rated from 1 (very much improved) to 7 (very much worse) with a higher score indicating a higher level of disease severity.
State-Trait Anxiety Inventory (State Component; STAI-State) | 1 day
  The State-Trait Anxiety Inventory (State component; STAI-State) is a self reported measure of subjective anxiety at the time of questionnaire completion. The range is 0-80 with a higher total score indicating a higher level of anxiety.

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - AFFIRM-1 Study Site, Encino, California
  - AFFIRM-1 Study Site, La Jolla, California
  - AFFIRM-1 Study Site, Los Angeles, California
  - AFFIRM-1 Study Site, Oceanside, California
  - AFFIRM-1 Study Site, San Diego, California
  - AFFIRM-1 Study Site, San Jose, California
  - AFFIRM-1 Study Site, Sherman Oaks, California
  - AFFIRM-1 Study Site, Temecula, California
  - AFFIRM-1 Study Site, Jacksonville, Florida
  - AFFIRM-1 Study Site, Lauderhill, Florida
  - AFFIRM-1 Study Site, Miami Lakes, Florida
  - AFFIRM-1 Study Site, Orlando, Florida
  - AFFIRM-1 Study Site, Tampa, Florida
  - AFFIRM-1 Study Site, Decatur, Georgia
  - AFFIRM-1 Study Site, Boston, Massachusetts
  - AFFIRM-1 Study Site, Princeton, New Jersey
  - AFFIRM-1 Study Site, Brooklyn, New York
  - AFFIRM-1 Study Site, Charlotte, North Carolina
  - AFFIRM-1 Study Site, Media, Pennsylvania
  - AFFIRM-1 Study Site, Austin, Texas

REFERENCES:
- See also: Study information and pre-screening portal for potential participants — https://theaffirm1study.com/